CLINICAL TRIAL: NCT00259194
Title: Observation and Prediction of Complications After Coronary Angiography
Acronym: OPKAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herning Hospital (Other)
Collaborators: The Medical Research Fund of the County of Ringkøbing (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OPKAT
Record Dates: First submitted 2005-11-28; First posted 2005-11-29 (Estimated); Last update posted 2009-06-11 (Estimated); Status verified 2009-06

CONDITIONS: Coronary Arteriosclerosis; Myocardial Ischemia
Keywords: Coronary angiography; Complications; Observation
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alternative Observation (Active Comparator): Moving in bed during observation after coronary angiography
  Interventions: Behavioral: Moving
- Standard Observation (Experimental): No moving in bed during observation after coronary angiography
  Interventions: Behavioral: No Moving

INTERVENTIONS:
Behavioral: Moving — The patients are allowed to lift their head, arms and legs during the 2 hours.
  Arms: Alternative Observation
Behavioral: No Moving — The patients are told not to move, to keep their legs and upper arms down and not to lift the head from the pillow in these 2 hours.
  Arms: Standard Observation

SUMMARY:
Coronary angiography via the femoral artery is regarded as a safe procedure, but bleeding complications are often seen. To avoid/reduce bleeding complications digital compression is applied in the area of puncture during approximately 20 minutes and the patient is in the investigators' department observed in bed for 2 hours. The investigators apply pressure over the puncture site using a sand bag in the first hour. The patients are told not to move, to keep their legs and upper arms down and not to lift the head from the pillow in these 2 hours (standard observation). In the present study the patients are randomized between standard observation and an alternative observation, where the patients are allowed to lift their head, arms and legs during the 2 hours, otherwise as standard observation.

The study has three aims:

1. To establish the incidence of bleeding complications:

   * Frequency of hematoma (> 5 cm)
   * Frequency of pseudoaneurysms
   * Frequency of bleeding demanding surgery
   * Frequency of bleeding demanding transfusion
2. Establish a model to predict in wich patient to expect a bleeding complication.
3. Assess if the alternative observation is associated with more bleeding complications compared to standard observation.

ELIGIBILITY:
Inclusion Criteria:

1. Coronary angiography by the femoral access, where the arterial lumen is reached.
2. Only attempted puncture at one side.
3. Age >= 18 years.

Exclusion Criteria:

1. Conditions that makes observation in the department impossible.
2. Dementia or other reasons to expect lack of compliance.
3. Previous participation in the project.
4. Implanted vascular prothesis at puncture site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2005-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Incidence of bleeding complications | 4 days
Model to predict bleeding complications | 4 days
Assess if lying still in bed the first 2 hours after angiography affect the incidence of bleeding complications | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Ole May, Dr.,Ph.D., Study Chair — Dept. of Med., Section of Cardiol., Herning Hospital, DK-7400 Herning
Locations (2):
- Denmark (2):
  - Coronary Angiography Laboratory, Herning
  - Dept. of Med., Sect. of Cardology, Herning Hospital, Herning

REFERENCES:
- [Result] May O, Schlosser H, Skytte L. A high blood pressure predicts bleeding complications and a longer hospital stay after elective coronary angiography using the femoral approach. J Interv Cardiol. 2009 Apr;22(2):175-8. doi: 10.1111/j.1540-8183.2009.00427.x. Epub 2009 Feb 24. PMID 19245381
- [Result] May O, Schlosser H, Skytte L. A randomized trial assessing the influence of lying still or being allowed to move in the observation period following coronary angiography using the femoral approach. J Interv Cardiol. 2008 Aug;21(4):347-9. doi: 10.1111/j.1540-8183.2008.00359.x. Epub 2008 May 29. PMID 18513345